CLINICAL TRIAL: NCT03182478
Title: Improving Skin Picking Treatment Using a Cognitive-Behavioral Protocol in Individual and Group Format: a Randomized Clinical Trial
Brief Title: Treating Skin Picking With Cognitive-Behavioral Protocol in Individual and Group Format.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Carolina Blaya Dreher, Carolina Blaya Dreher, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1185-5527
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Skin-Picking
Keywords: skin picking; SPD; Cognitive-Behavioral Therapy; CBT; Group treatment; Rothbaum protocol
MeSH Terms: conditions — Excoriation Disorder

STUDY DESIGN:
Intervention Model Description: Intervention with Rothbaum protocol adapted to skin picking disorder, in individual or group format, consisting of eight weekly sessions, each session during 45 minutes in individual format and 90 minutes in group format
Who Masked: Outcomes Assessor
Masking Description: Patients will be evaluated through scales applied before and after intervention by investigators that will be blinded about the intervention arm of the patient (individual or group format)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Treatment (Active Comparator): Intervention with the Rothbaum Protocol in individual format, with eight weekly sessions each one of 45 minutes, applied by a trained investigator. Session 1: Psychoeducation and self-monitoring. Session 2: habit reversal techniques. Session 3: muscle relaxation and diaphragmatic breathing. Session 4: stop the thought. Session 5: oriented internal dialogue. Session 6: cognitive techniques. Session 7: role-play. Session 8: relapse prevention
  Interventions: Behavioral: Rothbaum protocol in individual format
- Group Treatment (Active Comparator): Intervention with the Rothbaum Protocol in group format up to 10 patients, with eight weekly sessions each one of 90 minutes, applied by a trained investigator. Session 1: Psychoeducation and self-monitoring. Session 2: habit reversal techniques. Session 3: muscle relaxation and diaphragmatic breathing. Session 4: stop the thought. Session 5: oriented internal dialogue. Session 6: cognitive techniques. Session 7: role-play. Session 8: relapse prevention
  Interventions: Behavioral: Rothbaum protocol in group format

INTERVENTIONS:
Behavioral: Rothbaum protocol in individual format — 8-week 45 minute session Rothbaum CBT protocol adapted to Skin Picking, changing the focus on pulling hair to picking skin. Session 1: psychoeducation of the skin picking habit and how CBT works, patients initiate the self-monitoring of the habit. Session 2: techniques of habit reverse, adapted by having the skin as a target instead of the hair. The session 3: anxiety management using diaphragmatic breathing and muscle relaxation. Sessions 4 to 6: management of dysfunctional thoughts, using cognitive tools as the evidence analysis, reattribution of roles and gravity scale. Session 7: change of roles and role-playing, with patient playing the role of therapist, applying the Rothbaum Protocol to treat Skin Picking, so reviewing all the protocol techniques. Session 8: relapse prevention.
  Other Names: Cognitive-Behavioral Protocol
  Arms: Individual Treatment
Behavioral: Rothbaum protocol in group format — 8-week 90 minute session of Rothbaum CBT protocol adapted to Skin Picking, changing the focus on pulling hair to picking skin. Session 1: psychoeducation of the skin picking habit and how CBT works, patients initiate the self-monitoring of the habit. Session 2: techniques of habit reverse, adapted by having the skin as a target instead of the hair. The session 3: anxiety management using diaphragmatic breathing and muscle relaxation. Sessions 4 to 6: management of dysfunctional thoughts, using cognitive tools as the evidence analysis, reattribution of roles and gravity scale. Session 7: change of roles and role-playing, with patient playing the role of therapist, applying the Rothbaum Protocol to treat Skin Picking, so reviewing all the protocol techniques. Session 8: relapse prevention.
  Other Names: Cognitive-behavioral protocol
  Arms: Group Treatment

SUMMARY:
Skin Picking Disorder (SPD) affects 1.4-5.4% of the general population. It has a high association with anxiety and depressive symptoms. Only behavioral treatments demonstrated significant benefits compared with inactive control conditions, but with poor accessibility of this treatment to patients. Besides this, behavioral treatment does not address the associated anxious and depressive symptoms. Trichotillomania and SPD have co-occurrence rate greater than expected, indicating that can be part of the same disease spectrum. The Rothbaum Cognitive Behavioral Therapy(CBT) protocol is effective in treating trichotillomania. Based on the similarity of these diseases, this study uses the Rothbaum Protocol to treat SPD in individual and group format. We hypothesize that this protocol will be effective in treating SPD, anxiety and depression symptoms associated and also facilitate therapist training. Methods: A community sample of 40 participants with SPD will be randomly allocated to receive treatment with the Rothbaum Protocol individually or in group format. Patients with current psychotic disorder, suicide risk or mental disability will be excluded. Instruments measuring anxiety, depression and SPD severity will be applied in the baseline, after the intervention and after a 6 months follow-up. Motivation of patients to therapy will be evaluated at the baseline. The primary outcome will be the remission of symptoms evaluated by the overall clinical impression. The secondary outcomes will be the degree of improvement in anxiety, depression and SPD severity.

DETAILED DESCRIPTION:
Skin Picking Disorder (SPD) is a new diagnosis in the Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 and affects about 1.4% to 5.4% of the general population, increasing this prevalence to 7% to 30% in psychiatric patients. Despite the importance of this pathology, less than half of the patients with SPD seek treatment, only 53% receive the correct diagnosis and more than 57% are not satisfied with the treatment received. About 85% of patients think that professionals are not trained to treat SPD. Skin Picking Disorder occurs frequently with other mental disorders, with 13-48% of patients having major depressive disorder and 5-23% having anxiety disorders. The literature suggests that neither Selective Serotonin Reuptake Inhibitors (SSRIs) nor Lamotrigine are effective when compared to placebo in treating SPD, and only treatment with behavioral techniques are effective. However, studies using behavioral techniques do not address associated symptoms, as anxiety and depression.

Some studies found that the rate of co-occurrence of dermatillomania and trichotillomania is higher than expected, so it has been hypothesized that these disorders are part of the spectrum of a single pathology. It is known that the Rothbaum Protocol, a standardized treatment for Trichotillomania, is effective in treating this disorder, addressing also the management of anxiety and depressive symptoms, besides working with relapse prevention.

Thus, our study works with the hypothesis that the Rothbaum CBT Protocol can be effective in the treatment of dermatillomania, in both individual or group format. Having the same protocol to treat SPD and Trichotillomania might facilitate the patient access to treatment and the therapist training, and also might improve the SPD treatment in a long-term, by managing the relapse prevention.

Methods: this study is a thwo armed randomized controlled and single masked clinical trial. Participants with SPD according to DSM 5 will be included and randomly allocated in individual or group format of treatment with the Rothbaum CBT Protocol. The protocol will be adapted to SPD, changing the habit of pulling the hair to the habit of picking the skin. Symptoms of anxiety, depression and the SPD severity will be evaluated by specific instruments and by a photographic measurement before the intervention, after and in a 6 moths follow-up. The motivation of patient to the CBT will be measured at the baseline. Will be excluded patients with current psychotic disorder, suicide risk or mental disability.

The CBT protocol will consist of 8 weekly sessions, during 45 minutes in individual format and 90 minutes in group format, always applied by a trained therapist. This protocol includes psychoeducation, habit reversal techniques, anxiety management, change of disfunctional cognitive schemes and relapse prevention.

The primary outcome will be the remission of symptoms of SPD, assessed by the Clinical Global Impression scale. The secondary outcomes will be the improvement of depressive symptoms, anxiety and SPD symptoms assessed by the others instruments.

ELIGIBILITY:
Inclusion Criteria:

* Skin Picking diagnosis according to DSM 5 criteria

Exclusion Criteria:

* Current psychotic disorder
* Current suicide risk
* Intellectual disability

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Remission of symptoms | baseline, 8 weeks, 6 months
  Remission of Skin Picking symptoms, evaluated by the Clinical Global Impression Scale, with a score under or equal 2 considered remission.

SECONDARY OUTCOMES:
Improvement in anxious symptoms | baseline, 8 weeks, 6 months
  Mean Change From BaselineI in anxious symptoms assessed by the Hamilton Anxiety Scale
Improvement in depressive symptoms | baseline, 8 weeks, 6 months
  Mean Change From Baseline, assessed by the Beck Depression Inventory
Improvement in Skin Picking lesions | baseline, 8 weeks, 6 months
  Mean Change From Baseline, assessed by the photographic measurement
Improvement in Skin Picking life impact | baseline, 8 weeks, 6 months
  Mean Change From Baseline, assessed by the Skin Picking Impact Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Blaya Dreher, PhD, Study Director — Federal University of Health Science of Porto Alegre
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Pôrto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grant JE, Odlaug BL, Chamberlain SR, Keuthen NJ, Lochner C, Stein DJ. Skin picking disorder. Am J Psychiatry. 2012 Nov;169(11):1143-9. doi: 10.1176/appi.ajp.2012.12040508. PMID 23128921
- [Background] Snorrason I, Belleau EL, Woods DW. How related are hair pulling disorder (trichotillomania) and skin picking disorder? A review of evidence for comorbidity, similarities and shared etiology. Clin Psychol Rev. 2012 Nov;32(7):618-29. doi: 10.1016/j.cpr.2012.05.008. Epub 2012 Jul 20. PMID 22917741
- [Background] Hayes SL, Storch EA, Berlanga L. Skin picking behaviors: An examination of the prevalence and severity in a community sample. J Anxiety Disord. 2009 Apr;23(3):314-9. doi: 10.1016/j.janxdis.2009.01.008. Epub 2009 Jan 23. PMID 19223150
- [Background] Gupta MA, Gupta AK. Current concepts in psychodermatology. Curr Psychiatry Rep. 2014 Jun;16(6):449. doi: 10.1007/s11920-014-0449-9. PMID 24740235
- [Background] Tucker BT, Woods DW, Flessner CA, Franklin SA, Franklin ME. The Skin Picking Impact Project: phenomenology, interference, and treatment utilization of pathological skin picking in a population-based sample. J Anxiety Disord. 2011 Jan;25(1):88-95. doi: 10.1016/j.janxdis.2010.08.007. Epub 2010 Aug 13. PMID 20810239
- [Background] Keuthen NJ, Tung ES, Reese HE, Raikes J, Lee L, Mansueto CS. Getting the word out: cognitive-behavioral therapy for trichotillomania (hair-pulling disorder) and excoriation (skin-picking) disorder. Ann Clin Psychiatry. 2015 Feb;27(1):10-5. PMID 25696776
- [Background] Schuck K, Keijsers GP, Rinck M. The effects of brief cognitive-behaviour therapy for pathological skin picking: A randomized comparison to wait-list control. Behav Res Ther. 2011 Jan;49(1):11-7. doi: 10.1016/j.brat.2010.09.005. Epub 2010 Sep 22. PMID 20934685
- [Background] Selles RR, McGuire JF, Small BJ, Storch EA. A systematic review and meta-analysis of psychiatric treatments for excoriation (skin-picking) disorder. Gen Hosp Psychiatry. 2016 Jul-Aug;41:29-37. doi: 10.1016/j.genhosppsych.2016.04.001. Epub 2016 Apr 13. PMID 27143352
- [Derived] Xavier ACM, de Souza CMB, Flores LHF, Bermudez MB, Silva RMF, de Oliveira AC, Dreher CB. Skin picking treatment with the Rothbaum cognitive behavioral therapy protocol: a randomized clinical trial. Braz J Psychiatry. 2020 Sep-Oct;42(5):510-518. doi: 10.1590/1516-4446-2019-0636. PMID 32401873